CLINICAL TRIAL: NCT04532554
Title: The Impact of Growth Hormone in Obese Cases With Covid-19
Brief Title: Growth Hormone in Obese Cases With Covid-19
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: ClinAmygate (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR0015
Record Dates: First submitted 2020-08-24; First posted 2020-08-31 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Growth Hormone; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth hormone (Experimental): Recombinant GH will be used for those patients
  Interventions: Drug: Growth Hormone
- Placebo (Placebo Comparator): Saline will be used
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Growth Hormone — Recombinant growth hormone will be used
  Other Names: Recombinant growth hormone
  Arms: Growth hormone
Drug: Placebo — Saline injection with the same amount
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The use of growth hormone in obese cases with COVID-19 may help them to recover earlier.

DETAILED DESCRIPTION:
It is well known that lymphoid organs such the thymus, the spleen and peripheral blood produce growth hormone (GH) and GH receptor is expressed on different subpopulations of lymphocytes. Many in vitro and in animal studies demonstrate an important role of GH in immunoregulation. GH stimulates T and B cells proliferation and immunoglobulin synthesis, enhances the maturation of myeloid progenitor cells and is also able to modulate cytokine response.

The use of growth hormone in obese cases with COVID-19 may help them to recover earlier.

ELIGIBILITY:
Inclusion Criteria:

* Obese with BMI > 30

Exclusion Criteria:

* History of hypersensitivity to GH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-26 (Estimated); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Need for hospitalization | one to two weeks
  need to be hospitalized due to deterioration

SECONDARY OUTCOMES:
Time to recovery | one to four weeks
  Time to recovery from symptoms and signs
Percentage of reduction in CRP | one to two weeks
  Percentage of reduction in CRP
Percentage of reduction in LDH | one to two weeks
  Percentage of reduction in LDH
Percentage of reduction in Ferritin | one to two weeks
  Percentage of reduction in Ferritin
Time to recovery from leucopenia | one to two weeks
  Time to recovery from leucopenia

CONTACTS AND LOCATIONS:
Overall Officials: Emad R Issak, MD, Principal Investigator — Assalam Clinics
Locations (1):
- Asalam, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meazza C, Pagani S, Travaglino P, Bozzola M. Effect of growth hormone (GH) on the immune system. Pediatr Endocrinol Rev. 2004 Aug;1 Suppl 3:490-5. PMID 16444180
- See also: Effect of growth hormone (GH) on the immune system. — https://www.researchgate.net/publication/7329964_Effect_of_growth_hormone_GH_on_the_immune_system